CLINICAL TRIAL: NCT06999265
Title: Effect of Peripheral Neuromodulation on Vaginal Blood Flow
Brief Title: Effect of Peripheral Neuromodulation on Vaginal Blood Flow - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: International Society for the Study of Women's Sexual Health (Unknown); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Timothy Bruns, Associate Professor of Biomedical Engineering, Medical School, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00148746-b
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Female Sexual Dysfunction; Female Sexual Dysfunction Due to Physical Condition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tibial nerve stimulation, then genital nerve stimulation (Experimental): Participants in this arm received tibial nerve stimulation during their first study visit. Those who returned for the second study visit then received genital nerve stimulation. Film Clip Alternation will take place during both interventions.
  Interventions: Device: Transcutaneous electrical nerve stimulation - Tibial Nerve; Device: Transcutaneous electrical nerve stimulation - Genital Nerve; Behavioral: Neutral and Erotic Film Clip Alternation
- Genital nerve stimulation, then tibial nerve stimulation (Experimental): Participants in this arm received genital nerve stimulation during their first study visit. Those who returned for the second study visit then received tibial nerve stimulation. Film Clip Alternation will take place during both interventions.
  Interventions: Device: Transcutaneous electrical nerve stimulation - Tibial Nerve; Device: Transcutaneous electrical nerve stimulation - Genital Nerve; Behavioral: Neutral and Erotic Film Clip Alternation

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation - Tibial Nerve — Standard Transcutaneous electrical nerve stimulation (TENS) device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
Device: Transcutaneous electrical nerve stimulation - Genital Nerve — Standard Transcutaneous electrical nerve stimulation (TENS) device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
Behavioral: Neutral and Erotic Film Clip Alternation — During the testing period, participants will first view a 5-minute neutral film depicting nature scenes to allow blood flow levels to stabilize. This will be followed by a 10-minute period while the subject watches an erotic film clip for assessment of arousal responses without electrical stimulation. A 10-minute clip of the same neutral film will follow, to allow blood flow levels to return to baseline. Five minutes into this film, electrical stimulation will be resumed at the previously determined amplitude. Finally, the subject will view another 10-minute erotic film clip depicting similar sexually explicit material as the first while electrical stimulation remains on as the last sequence in the testing. Physiological arousal will be assessed with a vaginal photoplethysmography probe, yielding vaginal pulse amplitude (VPA) for analysis. Subjective arousal will be assessed with a subjective arousal questionnaire.

SUMMARY:
The overall purpose of this research is to improve sexual function in women with sexual dysfunction. The goal of this study is to see if either of two nerve stimulation interventions cause a short-term change in vaginal blood flow. The effect of this intervention will be compared between women who have neurogenic (spinal cord injury) or non-neurogenic dysfunction and healthy women, to reveal mechanisms underlying neural control over vaginal blood flow.

DETAILED DESCRIPTION:
This study will explore the short-term effect of tibial and genital stimulation on vaginal blood flow in healthy women, non-neurogenic women with female sexual dysfunction (FSD), and women with both FSD and spinal cord injuries (SCI). To potentially amplify any stimulation effects, this study will incorporate the use of sexually explicit films, a method that is standard in sexual function studies.

ELIGIBILITY:
Inclusion Criteria:

All Participants

* All participants will need internet access to complete the initial surveys and the diaries.

Non-dysfunction participants

* Adult (over 18 years old) cis-gender female
* Neurologically stable
* Sexually active at least once per month
* Able to understand consent and communicate effectively with research team

Non-SCI dysfunction participants

* Adult (over 18 years old) cis-gender female
* Neurologically stable
* Sexually active at least once per month
* Sexual dysfunction, per short-form Female Sexual Function Index (FSFI) score below 19
* Lubrication difficulties, per short-form FSFI lubrication subdomain score below or equal to 3
* Able to understand consent and communicate effectively with research team

Spinal cord injured participants

* Adult (over 18 years old) cis-gender female
* Clinically diagnosed spinal cord injury (Impairment score A-B) at vertebral level within C6-T10 at least six months prior or clinically diagnosed spinal cord injury (Impairment score C) at vertebral level within C4-T10 at least six months prior
* Nominally sexually active, but at minimum interest in sexual pleasure even if fully self-induced
* Sexual dysfunction, per short-form FSFI score below 19
* Able to understand consent and communicate effectively with research team

Exclusion Criteria:

Non-dysfunction participants:

* Male
* Pregnancy or planning to become pregnant during study period
* Sexual dysfunction, per short-form FSFI score below 19
* Lubrication difficulties, per short-form FSFI lubrication subdomain score below or equal to 4, or per investigator's discretion
* Clinically diagnosed bladder dysfunction, pelvic pain, or other pelvic organ symptoms
* Suspected or diagnosed epilepsy
* Active infection or active pressure sores in the perineal region
* Implanted pacemaker or defibrillator
* Currently has or tested positive in the last 14 days for COVID-19 or is symptomatic for COVID-19

Non-SCI dysfunction participants:

* Male
* Pregnancy or planning to become pregnant during study period
* Clinically diagnosed bladder dysfunction, pelvic pain, or other pelvic organ symptoms
* Suspected or diagnosed epilepsy
* Active infection or active pressure sores in the perineal region
* Implanted pacemaker or defibrillator
* Currently has or tested positive in the last 14 days for COVID-19 or is symptomatic for COVID-19

Spinal cord injured participants:

* Male
* Spinal cord injury at or above C5 level (C1-C5) if Impairment score A or B, or spinal cord injury at or above C3 level (C1-C3) if Impairment score C
* Spinal cord injury below T10 vertebral level or reflexes not preserved
* Acute worsening in motor or sensory function in the last month
* Suspected or diagnosed epilepsy
* Pregnancy or planning to become pregnant during study period
* Active infection or active pressure sores in the perineal region
* Implanted pacemaker or defibrillator
* Currently has or tested positive in the last 14 days for COVID-19 or is symptomatic for COVID-19

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only cisgendered females were eligible for this study
Enrollment: 15 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bruns, Ph.D, Principal Investigator — University of Michigan; Priyanka Gupta, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tibial Nerve Stimulation, Then Genital Nerve Stimulation: Participants in this arm received tibial nerve stimulation during their first study visit. Those who returned for the second study visit then received genital nerve stimulation. Film Clip Alternation will take place during both interventions.
  Transcutaneous electrical nerve stimulation (TENS) - Tibial Nerve: TENS device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
  Transcutaneous electrical nerve stimulation (TENS) - Genital Nerve: TENS device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
  Neutral and Erotic Film Clip Alternation: During the testing period, participants will first view a 5-minute neutral film depicting nature scenes to allow blood flow levels to stabilize. This will be followed by a 10-minute period while the subject watches an erotic film clip for assessment of arousal responses without electrical stimulation. A 10-minute clip of the same neutral film will follow, to allow blood flow levels to return to baseline. Five minutes into this film, electrical stimulation will be resumed at the previously determined amplitude. Finally, the subject will view another 10-minute erotic film clip depicting similar sexually explicit material as the first while electrical stimulation remains on as the last sequence in the testing.
- Genital Nerve Stimulation, Then Tibial Nerve Stimulation: Participants in this arm received genital nerve stimulation during their first study visit. Those who returned for the second study visit then received tibial nerve stimulation. Film Clip Alternation will take place during both interventions.
  Transcutaneous electrical nerve stimulation (TENS) - Tibial Nerve: TENS device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
  Transcutaneous electrical nerve stimulation (TENS) - Genital Nerve: TENS device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
  Neutral and Erotic Film Clip Alternation: During the testing period, participants will first view a 5-minute neutral film depicting nature scenes to allow blood flow levels to stabilize. This will be followed by a 10-minute period while the subject watches an erotic film clip for assessment of arousal responses without electrical stimulation. A 10-minute clip of the same neutral film will follow, to allow blood flow levels to return to baseline. Five minutes into this film, electrical stimulation will be resumed at the previously determined amplitude. Finally, the subject will view another 10-minute erotic film clip depicting similar sexually explicit material as the first while electrical stimulation remains on as the last sequence in the testing.
Period: Overall Study
Arm/Group | Tibial Nerve Stimulation, Then Genital Nerve Stimulation | Genital Nerve Stimulation, Then Tibial Nerve Stimulation
Started (First treatment option (randomized tibial or genital)) | 10 | 5
Completed (Second treatment option (opposite from first)) | 9 | 4
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tibial Nerve Stimulation, Then Genital Nerve Stimulation | Genital Nerve Stimulation, Then Tibial Nerve Stimulation | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.7) | 35.6 (10.7) | 37.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 6 | 3 | 9
  Multiracial | 0 | 0 | 0
  Asian/Pacific Islander | 3 | 1 | 4
  Black/African American | 1 | 1 | 2
  Native American/American Indian/Alaskan Native | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 5 | 15
Baseline Vaginal Pulse Amplitude (VPA) [Mean (Standard Deviation); unit: mV] — Vaginal Pulse Amplitude (VPA) is measured with a vaginal photoplethysmograph probe, which provides a measure of local blood flow in a relative scale using mV. The baseline VPA measure for each participant was determined as the mean VPA during the baseline period.
  The Outcome measure was calculated as mean baseline of the total participants, regardless of which order they were administered the treatment. One participant in the Tibial Nerve First arm did not receive the Genital Nerve treatment. One participant in the Genital Nerve First arm did not receive the Tibial Nerve treatment. Population: Measure Description: Outcome measure was calculated as baseline of the total participants, regardless of which order they were administered the treatment. One participant in the Tibial Nerve First arm did not receive the Genital Nerve treatment. One participant in the Genital Nerve First arm did not receive the Tibial Nerve treatment.
  mV
    Tibial Nerve VPA Baseline: number analyzed (Participants) | 10 | 4 | 14
    Tibial Nerve VPA Baseline | 20.6 (10.1) | 12.8 (14.0) | 18.3 (11.4)
    Genital Nerve VPA Baseline: number analyzed (Participants) | 9 | 5 | 14
    Genital Nerve VPA Baseline | 21.5 (16.5) | 17.6 (15.0) | 20.1 (15.5)
Baseline Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Outcome measure was calculated as baseline of the total participants, regardless of which order they were administered the treatment. One participant in the Tibial Nerve First arm did not receive the Genital Nerve treatment. One participant in the Genital Nerve First arm did not receive the Tibial Nerve treatment. Population: Measure Description: Outcome measure was calculated as baseline of the total participants, regardless of which order they were administered the treatment. One participant in the Tibial Nerve First arm did not receive the Genital Nerve treatment. One participant in the Genital Nerve First arm did not receive the Tibial Nerve treatment.
  beats per minute
    Tibial Nerve Stimulation Baseline: number analyzed (Participants) | 10 | 4 | 14
    Tibial Nerve Stimulation Baseline | 69.3 (10.9) | 63.7 (4.9) | 67.7 (9.8)
    Genital Nerve Stimulation Baseline: number analyzed (Participants) | 9 | 5 | 14
    Genital Nerve Stimulation Baseline | 67.3 (7.1) | 68.8 (8.7) | 67.8 (7.4)
Baseline Mean Arterial Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Measure Description: Outcome measure was calculated as baseline of the total participants, regardless of which order they were administered the treatment. One participant in the Tibial Nerve First arm did not receive the Genital Nerve treatment. One participant in the Genital Nerve First arm did not receive the Tibial Nerve treatment. Population: Measure Description: Outcome measure was calculated as baseline of the total participants, regardless of which order they were administered the treatment. One participant in the Tibial Nerve First arm did not receive the Genital Nerve treatment. One participant in the Genital Nerve First arm did not receive the Tibial Nerve treatment.
  mm Hg
    Tibial Nerve Stimulation Baseline: number analyzed (Participants) | 10 | 4 | 14
    Tibial Nerve Stimulation Baseline | 81.8 (4.0) | 79.3 (4.1) | 81.1 (4.0)
    Genital Nerve Stimulation Baseline: number analyzed (Participants) | 9 | 5 | 14
    Genital Nerve Stimulation Baseline | 85.2 (8.8) | 82.6 (6.4) | 84.2 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Change in Vaginal Pulse Amplitude (VPA) From the Average Baseline Value
Description: VPA will be measured by a vaginal plethysmography transducer that is placed in the vagina to measure changes in blood flow during the full study session.
  Overall treatment sequence:
  baseline (nature) video erotic video 1 (no treatment = "control") baseline nature video (treatment on in middle) erotic video 2 (treatment)
  The average VPA value during the baseline period will be determined. The maximum percent change in VPA during each relevant sequence as compared to the average baseline VPA will be determined for each participant.
Time Frame: Up to five months
Population: Analysis population is all participants who received the designated treatment, regardless of which treatment they received first or if they continued to the second treatment.
Measure: Mean (Standard Deviation); unit: percent change of VPA
Groups:
- Tibial Nerve Stimulation: Participants received tibial nerve stimulation and Film Clip Alternation.
  Transcutaneous electrical nerve stimulation (TENS) - Tibial Nerve: TENS device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
  Neutral and Erotic Film Clip Alternation: During the testing period, participants will first view a 5-minute neutral film depicting nature scenes to allow blood flow levels to stabilize. This will be followed by a 10-minute period while the subject watches an erotic film clip for assessment of arousal responses without electrical stimulation. A 10-minute clip of the same neutral film will follow, to allow blood flow levels to return to baseline. Five minutes into this film, electrical stimulation will be resumed at the previously determined amplitude. Finally, the subject will view another 10-minute erotic film clip depicting similar sexually explicit material as the first while electrical stimulation remains on as the last sequence in the testing.
- Genital Nerve Stimulation: Participants received genital nerve stimulation and Film Clip Alternation.
  Transcutaneous electrical nerve stimulation (TENS) - Genital Nerve: TENS device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
  Neutral and Erotic Film Clip Alternation: During the testing period, participants will first view a 5-minute neutral film depicting nature scenes to allow blood flow levels to stabilize. This will be followed by a 10-minute period while the subject watches an erotic film clip for assessment of arousal responses without electrical stimulation. A 10-minute clip of the same neutral film will follow, to allow blood flow levels to return to baseline. Five minutes into this film, electrical stimulation will be resumed at the previously determined amplitude. Finally, the subject will view another 10-minute erotic film clip depicting similar sexually explicit material as the first while electrical stimulation remains on as the last sequence in the testing.
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
Number analyzed (Participants) | 14 | 14
percent change of VPA
  baseline to end of first erotic video | 119.8 (107.4) | 94.3 (76.2)
  baseline to end of second erotic video | 135.4 (153.9) | 113.5 (92.3)
  end of first video to end of second erotic video | 9.9 (45.2) | 15.0 (37.9)

2. Secondary Outcome: Percent Change in Heart Rate From Baseline
Description: A heart rate monitor (e.g. electrocardiogram or pulse oximetry) will be placed on the participant's arm, hand, or chest (as is appropriate per monitor) to measure the heart rate in beats per minute (bpm).
  The average heart rate in bpm during the baseline video will be determined. The average percent change in heart rate during each test sequence as compared to the average baseline heart rate will be determined.
Time Frame: Up to five months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change of heart rate
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
Number analyzed (Participants) | 14 | 14
percent change of heart rate
  baseline to end of first erotic video | 2.4 (6.1) | 0.8 (6.9)
  baseline to end of second erotic video | -0.5 (6.6) | 2.8 (5.7)
  end of first video to end of second erotic video | -2.8 (5.5) | 2.1 (5.0)

3. Secondary Outcome: Percent Change in Mean Arterial Blood Pressure From Baseline
Description: A blood pressure monitor will be placed on the participant's arm, hand, or chest (as is appropriate per monitor) to monitor off-target autonomic responses.
  The mean arterial blood pressure in millimeters of mercury (mm Hg) will be calculated for a period as the diastolic pressure plus 1/3 times the difference between the systolic pressure and the diastolic pressure, following standard practice.
  The average mean arterial blood pressure will be determined for the baseline period.
  The percent change in average mean arterial blood pressure with respect to the baseline period will be determined for each test sequence.
Time Frame: Up to five months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change of mean arterial blood pr
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
Number analyzed (Participants) | 14 | 14
percent change of mean arterial blood pr
  baseline to end of first erotic video | 1.8 (5.5) | 1.9 (4.6)
  baseline to end of second erotic video | 2.1 (5.6) | 3.4 (7.0)
  end of first video to end of second erotic video | 0.3 (3.3) | 1.5 (4.3)

4. Secondary Outcome: Change in Subjective Arousal From Baseline
Description: Subjective arousal will be evaluated by participants using a five point Likert scale, where 1 being no arousal and 5 being greatest arousal. Survey will be presented to patients between every video transition (a total of 4 times). Data is presented as averages per video transition point.
Time Frame: Up to five months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline, before video 1 (Survey 1) | 1.1 (0.4) | 1.4 (0.6)
  After video 1 (Survey 2) | 3.5 (0.9) | 3.4 (0.5)
  Before video 2 (Survey 3) | 1.4 (0.6) | 1.6 (0.8)
  After video 2 (Survey 4) | 3.9 (1.1) | 4.0 (0.5)

ADVERSE EVENTS:
Time Frame: Up to five months
Description: Participants were monitored for AEs during treatments and were given contact information for the study team so they could report AEs that happened after the treatments.
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT06999265/Prot_SAP_000.pdf